CLINICAL TRIAL: NCT01100411
Title: Changes in Invitro and ex Vivo Lens Metrology With Experienced Daily Wear Contact Lens Wearers
Brief Title: Changes in Invitro and ex Vivo Lens Metrology With Daily Wear Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M-10-01
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2011-11

CONDITIONS: Myopia
Keywords: Contact lenses, myopia, lens geometry
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Air Optix Aqua (Active Comparator): Contact lens material: Lotrafilcon A
  Interventions: Device: Air Optix Aqua
- Biofinity (Active Comparator): Contact lens material: Comfilcon A
  Interventions: Device: Biofinity
- Proclear (Active Comparator): Contact lens material: Omafilcon A
  Interventions: Device: Proclear
- Acuvue Oasys (Active Comparator): Contact lens material: Senofilcon A
  Interventions: Device: Acuvue Oasys
- Acuvue 2 (Active Comparator): Contact lens material: Etafilcon A
  Interventions: Device: Acuvue 2
- Purevision (Active Comparator): Contact lens material: Balafilcon A
  Interventions: Device: Purevision

INTERVENTIONS:
Device: Air Optix Aqua — Contact lens material: Lotrafilcon A
  Other Names: Air Optix
  Arms: Air Optix Aqua
Device: Biofinity — Contact lens material: Comfilcon A
  Other Names: CV Biofininty
  Arms: Biofinity
Device: Proclear — Contact lens material: Omafilcon A
  Other Names: Proclear Compatibles
  Arms: Proclear
Device: Acuvue Oasys — Contact lens material: Senofilcon A
  Other Names: Oasys
  Arms: Acuvue Oasys
Device: Acuvue 2 — Contact lens material: Etafilcon A
  Other Names: AV 2
  Arms: Acuvue 2
Device: Purevision — Contact lens material: Balafilcon A
  Other Names: PV
  Arms: Purevision

SUMMARY:
The purpose of this study is to evaluate changes in contact lens geometry after lens wear

DETAILED DESCRIPTION:
The purpose of this study is to evaluate changes invitro and ex vivo in contact lens geometry in daily lens wear

ELIGIBILITY:
Inclusion Criteria:

* • Able to read and comprehend English and give informed consent as demonstrated by signing a record of informed consent;

  * Be at least 18 years old;
  * Willing to comply with the wearing and clinical trial visit schedule as directed by the investigator;
  * Have ocular health findings considered to be "normal" and which would not prevent the participant from safely wearing contact lenses;
  * Has vision correctable to at least 6/12 (20/40) or better at distance in each eye with contact lenses;
  * Be experienced at wearing contact lenses.

Exclusion Criteria:

* • Any pre-existing ocular irritation, injury or condition (including keratoconus and herpes keratitis) of the cornea, conjunctiva or eyelids that would preclude contact lens fitting and safe wearing of contact lenses;

  * Any systemic disease that adversely affects ocular health
  * An active corneal infection or any active ocular disease that would affect wearing of contact lenses;
  * Use of any topical ocular medication during trial with the exception of saline drops ;
  * Use of or a need for any systemic medication or topical medications which may alter normal ocular findings/are known to affect a participant's ocular health/physiology or contact lens performance
  * Eye surgery within 12 weeks immediately prior to enrolment for this trial;
  * Previous corneal refractive surgery;
  * Contraindications to contact lens wear;
  * Participated or currently enrolled in another clinical trial that may have affected vision or ocular physiology within the previous 2 weeks;
  * Be pregnant (formal testing of pregnancy is not required. A participant's verbal report is sufficient);
  * Worn soft contact lenses 2 calendar days or rigid gas permeable/ orthokeratology lenses 7 calendar days prior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Lens Geometry | 1 week

SECONDARY OUTCOMES:
Corneal Shape | 1 week
Conjunctival Staining | 1 week
  The conjunctival staining

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Call Center, Study Chair — Alcon Research
Locations (1):
- Institute for Eye Research, Sydney, New South Wales, Australia